CLINICAL TRIAL: NCT01395186
Title: Varicocelectomy To Treat Pain, Predictors Of Success : A Prospective Study
Brief Title: Varicocelectomy To Treat Pain, Predictors Of Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: mansoura university, mansoura university
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Varicocelectomy To Treat Pain,
Record Dates: First submitted 2011-07-11; First posted 2011-07-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2009-04

CONDITIONS: Pain
Keywords: varicocele; pain
MeSH Terms: conditions — Pain; Varicocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- varicocelectomy (Other): varicocelectomy for patients complaining of pain
  Interventions: Procedure: varicocelectomy

INTERVENTIONS:
Procedure: varicocelectomy — varicocelectomy for painful varicocele
  Other Names: varicocelctomy

SUMMARY:
there are many studies studying the effectiveness of surgical treatment in patients treated for infertility, but only a few reporting the results of varicocelectomy done for pain. This study attempted to examine the success rate of varicocele ligation when performed for the treatment of pain and to evaluate all the predictor factors that may affect the pain resolve

DETAILED DESCRIPTION:
varicocelectomy for patients complaining of pain and studying the effectiveness and all predictors that can affect the degree of response

ELIGIBILITY:
Inclusion Criteria:

* painful varicocele after failure of medical therapy

Exclusion Criteria:

* responders to medical therapy

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
pain resolve after varicocelectomy | 3 months foloow up
  degree of pain resolve after varicocelectomy

SECONDARY OUTCOMES:
semen parameters | 6 months
  count,motility, morphology based on WHO 1995

CONTACTS AND LOCATIONS:
Overall Officials: ramadan ellithy, md, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt